CLINICAL TRIAL: NCT04045899
Title: "A Randomized Controlled Study Comparing ProSeal Laryngeal Mask Airway, Air-Q LMA and Ambu AuraGain in Mechanically Ventilated Patients"
Brief Title: Comparison Between Three Supraglottic Airway Devices ProSeal Laryngeal Mask Airway, Air-Q LMA and Ambu AuraGain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr.Mahak Mehta (Other)
Responsible Party: Sponsor-Investigator, Dr.Mahak Mehta, POST GRADUATE STUDENT, Government Medical College, Haldwani
Organization: Government Medical College, Haldwani (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 328/GMC/IEC/2016/Reg.No.280
Record Dates: First submitted 2019-03-12; First posted 2019-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Proseal LMA vs Air-Q LMA vs Ambu AurGain LMA
Keywords: Comparison of device

STUDY DESIGN:
Intervention Model Description: Methods:This prospective, randomised, single-blind study was conducted on 150 American Society of Anesthesiologists physical status I-II, randomly allocated into 3 groups, undergoing elective surgical procedures under general anaesthesia.PLMATM, Air-Q® and Ambu AuraGainTM appropriate for weight or/and height was inserted.Primary outcome measure was insertion time.Airway sealing pressure,ease of insertion, number of attempts,overall success rate, glottis view,number of attempts of gastric tube placement , hemodynamic parameters and complications were also recorded.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ProSeal Laryngeal Mask Airway Group (Active Comparator): ProSeal LMA was inserted in 50 patients
  Interventions: Device: Proseal LMA
- Air-Q LMA Group (Experimental): Air-Q LMA was inserted in 50 patients
  Interventions: Device: Air-Q LMA
- Ambu AuraGain LMA Group (Experimental): Ambu AuraGain was inserted in 50 patients
  Interventions: Device: Ambu AuraGain LMA

INTERVENTIONS:
Device: Proseal LMA — The Proseal Laryngeal Mask Airway (p-LMA) has a dual cuff modified to provide better sealing, and a drainage tube for gastric tube insertion. These features attribute in increasing the safety of the p-LMA when used with positive pressure ventilation.
  Arms: ProSeal Laryngeal Mask Airway Group
Device: Air-Q LMA — Air-Q LMA has a self-pressurizing cuff which inflates to adequate pressure during positive pressure ventilation thus eliminating the adverse effects of cuff over inflation associated with the use of Supraglottic airway device with an inflatable cuff.
  Arms: Air-Q LMA Group
Device: Ambu AuraGain LMA — The AmbuAuraGain™ is a disposable, preformed second generation SAD, anatomically curved with integrated gastric access and intubation capability, taking patient safety and airway management efficiency to a new level.
  Arms: Ambu AuraGain LMA Group

SUMMARY:
The present study entitled, "A Randomized Controlled Study Comparing ProSeal Laryngeal Mask Airway, Air-Q LMA and Ambu AuraGain in mechanically ventilated patients." was conducted in during the period Nov 2016 - Aug 2018.

The Aim of the study was to compare the clinical performance of ProSeal-LMA (P-LMA) ,Air-Q and Ambu AuraGain in terms of efficacy and safety in anaesthetized and paralyzed patients on mechanical ventilation undergoing elective surgical procedures.

Objective was to study the three supraglottic devices with respect to following parameters:-number of insertion attempts and overall success rate, ease of insertion of device, time taken for placement of device, airway sealing pressure, glottic view, number of attempts of gastric tube placement, hemodynamic parameters: heart rate and mean arterial pressure: pre-insertion and 0,1,3,5 and 10 minutes post insertion and complications noted if any: blood staining of device and tongue, lip and dental trauma, laryngospasm ,sore throat, dysphagia, hoarseness of voice.

It was a randomized prospective single blind comparative study comprised of 150 ASA I - II patients, aged 18-65 years of either sex who weighed between 40 to 60 kg scheduled for elective surgical procedure of duration not more than 90 mins. After a thorough pre-anaesthetic check-up, informed written consent was obtained and the patients were randomized into 3 groups of 50 patients each as Group P(Proseal), Group Q (Air Q) and Group A (AuraGain) by computer generated randomization sequence.

DETAILED DESCRIPTION:
In this study PLMA, Air-Q® and Ambu AuraGain were compared undergoing elective surgeries under general anaesthesia. Primary outcome measure was insertion time. Airway sealing pressure,ease of insertion, number of attempts,overall success rate, glottis view,number of attempts of gastric tube placement , hemodynamic parameters and complications were also compared.

After approval from the institutional ethical committee, 150 patients were studied in a randomised prospective study, designed to compare PLMA , Air-Q® and Ambu AuraGain .The period of the study was from nov 2016 to aug 2018. This study was conducted according to Good Clinical Practice standards and the Helsinki Declaration.

The American Society of Anesthesiologists (ASA) physical status I and II patients, between 18-65 years of age, weighing from 40 to 60 kg of either sex, undergoing elective surgical procedures of duration not more than 90 minutes were selected for the study. The exclusion criteria included patients with anticipated difficult airway (mouth opening of <2 finger, Mallampati Score 4, limited neck extension, history of previous difficult intubation), upper respiratory tract infections,airway related conditions such as trismus, trauma or mass, cervical spine disease, obese with body mass index (BMI) ≥25kg/m2 ,pregnant females, patients at risk of aspiration (full stomach, hiatus hernia, gastro-oesophageal reflux disease, emergency surgery)and laparoscopic surgeries. Neck movement was assessed as Class: I-No reduction in movement, II-1/3rd reduction, III-2/3rd reduction, IV-Complete reduction.

Following detailed pre-anaesthetic check-up, informed written consent was obtained from all patients fulfilling the required criteria.Patients were randomly allocated into three groups namely Group P(ProSeal,n=50) ,Group Q (Air-Q®, n = 50) and Group A (AuraGain™, n = 50) using computer-generated randomisation sequence. Participants were assigned to specific groups by the operating room nurse in charge.

After attaching the standard monitors(ASA recommended), patients were pre-medicated with injection midazolam 0.05 mg/kg, glycopyrrolate 0.2 mg, dexamethasone 4 mg and nalbuphine 0.02mg/kg intravenously. All patients were pre-oxygenated for 3 min, and anaesthesia was induced with injection propofol 2 mg/kg. Injection vecuronium 0.1 mg/kg was given for neuromuscular blockade.

PLMA or Air-Q® or AuraGain™ appropriate for weight or/and height was inserted as per the manufacturers guidelines.After successful insertion, the cuff was inflated with air according to the size and type of LMA as per manufacturers guidelines, to prevent audible and palpable air leak. An effective airway was confirmed by bilateral symmetrical chest expansion on manual ventilation, auscultation of breath sounds, square waveform on capnography. Devices were fixed with adhesive tape applied to the maxilla on one side of the patient's face and passed over and under the tube in a single loop before fixing to the opposite maxilla.

Anaesthesia was maintained with oxygen, nitrous oxide and isoflurane and intermittent positive pressure ventilation. Haemodynamic parameters[heart rate(HR), mean arterial pressure(MAP)]were monitored before and after the insertion of the device. A lubricated gastric tube was placed in the stomach through the gastric channel. At the end of surgical procedure, anaesthesia was discontinued and residual neuromuscular blockade reversed with injection neostigmine and glycopyrrolate, followed by device removal. Complication if any was noted.

Insertion time, number of insertion attempts, overall success rate, ease of insertion, airway sealing pressure, glottis view, number of attempts of gastric tube insertion, hemodynamic parameters (HR and MAP) preinduction, induction and 1,3,5 and 10mins post induction and complications were noted. One attempt was defined as insertion of the LMA between the teeth until the LMA will be deemed to be correctly placed and its cuff will be properly inflated. In case of insertion attempts, maximum of three attempts were allowed. An attempt was considered unsuccessful, if there was failure to negotiate the device beyond oropharynx, significant leak present (both audible and auscultatory) or inadequate ventilation with EtCO2>45 mmHg. Failure of a device was defined as three unsuccessful insertion attempts or inadequate ventilation. After failure of three attempts, intubation was performed using conventional rigid laryngoscopy and case was recorded as failed and also deleted from the study. The ease of insertion of device based on Visual Analogue Scale(VAS) was recorded.0 was considered the easiest insertion of device and 10 being the most difficult insertion.Insertion time was defined as time interval (in seconds) elapsed from insertion of LMA between the dental arches until the confirmation of successful ventilation determined by chest wall movement, auscultation of breath sounds and square wave capnographic curves and no oropharyngeal leak with peak airway pressure ≥ 20cmH2O, which was recorded by an independent observer.The airway sealing pressure was measured by closing the expiratory valve of the circle system at a fixed gas flow of 3 L/min and recording the airway pressure at which equilibrium is reached. At this stage, a leak at mouth and stomach was ascertained. Glottic viewing was assessed by insertion of the fibreoptic bronchoscope through the airway channel of the respective LMA.A maximum of two attempts were allowed for gastric tube placement. Its correct placement was confirmed by injection of air and epigastric auscultation or aspiration of gastric contents. Failure was defined as inability to advance the orogastric tube into the stomach within two attempts. Blood staining of the device and tongue, lip or dental trauma was noted. Incidence of laryngospasm or hypoxia (defined as oxygen saturation <92%), if any, in intra-operative period was noted and managed accordingly. In post-operative period, an investigator blinded to study asked the patients about the signs of sore throat, dysphagia and hoarseness of voice. Incidence of hoarseness and sore throat, whether present or absent, were enquired in 24 h post-operatively.

The primary outcome measure of the study was insertion time. Based on a previous study investigators found mean insertion time in PLMA group was 23.43 seconds and SD of 3.54. Based on that, taking alpha 0.05, β =0.90 and 25% difference between the means as significant, investigators calculated 47 patients were required in each group; hence, the sample size was increased to 50 patients each.

The data were recorded in a Microsoft Excel Spreadsheet and analysed using SPSS statistics software version 24 (IBM SPSS Inc., Chicago, IL, USA). Continuous numerical variables were presented as mean (standard deviation) and intergroup differences were compared using one-way analysis of variance with post hoc correction. Categorical variables were presented as ratio or as n (%) and inter-group differences were compared using Kruskall-Wallis test. The P< 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria: • American Society of Anaesthesiologists (ASA) class I/II.

* Age 18-65 years of either sex.
* Weight between 40-60 kg of either sex.
* Elective Surgical procedures of duration not more than 90 minutes with no need for endotracheal intubation.

Exclusion Criteria:

* • Patients with anticipated difficult airway(Mouth opening of <2 finger, Mallampati class 4,limited neck extension, history of previous difficult intubation).

  * Restricted mouth opening
  * Pregnant females
  * Cervical spine disease
  * Obese with body mass index ≥25kg/m2.
  * Patients with upper respiratory tract infections.
  * Patients at the risk of gastroesophageal regurgitation (eg hiatus hernia,sepsis, Diabetes Mellitus,obesity,pregnancy or a history of upper gastrointestinal surgery)
  * Laparoscopic surgeries
  * Patients with airway related conditions such as trismus,trauma or mass.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Insertion Time of device measured in seconds | 10 minutes
  Time of insertion:
  The time interval(seconds) elapsed from insertion of SAD between the dental arches until the confirmation of successful ventilation determined by chest wall movement,auscultation of breath sounds and square wave capnographic curves and no oropharyngeal leak with peak airway pressure >/= 20 cm of H2O.The time will be measured with the help of stop watch.

SECONDARY OUTCOMES:
Number of attempts of insertion of device | 15 minutes
  Attempt will be defined as insertion of the LMA between the teeth until the LMA will be deemed to be correctly placed and its cuff will be properly inflated.
  A maximum of three attempts will be allowed. An attempt will be considered unsuccessful if -
  * Failure to negotiate beyond oropharynx.
  * Significant Leak present (both audible and auscultatory)
  * Inadequate ventilation to be confirmed by Et-CO2 >45 mmHg. Failure of a device is identified as three unsuccessful insertion attempts or inadequate ventilation.
  After failure of three attempts intubation will be performed using conventional rigid laryngoscopy and case will be recorded as failed.
Ease of insertion of device measured via VISUAL ANALOGUE SCALE | 15 minutes
  The ease of insertion of device based on VISUAL ANALOGUE SCALE will be recorded.(0=easiest insertion of device,10=most difficult insertion)
Airway Sealing Pressure of device measured in mmHg | 15 minutes
  The airway sealing pressure is measured at cuff pressure of 60 cmH2O by closing the expiratory valve of the circle system at a fixed gas flow of 3L/min and recording the airway pressure at which equilibrium is reached. At this stage a leak at mouth and stomach is ascertained.
Glottic View through the device measured in % | 10 minutes
  Glottic viewing will be assessed by insertion of the fibreoptic bronchoscope through the airway channel of the respective SGA devices.
Number of attempts of gastric tube placement | 20 minutes
  A maximum of two attempts were allowed for gastric tube placement. Its correct placement confirmed by injection of air and epigastric auscultation or aspiration of gastric contents. Failure was defined as inability to advance the orogastric tube into the stomach within two attempts.
Complications | 2hours
  * Note for any Blood staining of the device and tongue, lip and dental trauma.
  * Incidence of Laryngospasm in intra operative period will be noted and managed accordingly.
  * Sore Throat, Dysphagia and Hoarseness of voice.
  In post-operative period an investigator blinded to study, will ask the patients about the signs of:
  1. Sore throat
  2. Dysphagia.
  3. Hoarseness of voice.
  Sore throat will be assessed to a score of 0-3:
  0: No pain
  1. Mild pain
  2. moderate pain
  3. Severe pain
  Dysphagia and hoarseness in voice was assessed on a score of 0-1:
  0: Absent
  1: Present
Mean Blood Pressure measured in mmHg | 30 minutes
  Preinsertion ,0,1,3,5 and 10 minutes post insertion
Heart Rate measured in beats per minute | 30 minutes
  Preinsertion ,0,1,3,5 and 10 minutes post insertion

CONTACTS AND LOCATIONS:
Overall Officials: MAHAK MEHTA, MD, Principal Investigator — M.B.B.S M.D Anaesthesia GMC Haldwani(Nainital)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Sood J. Laryngeal mask airway and its variants. Indian J Anaesth. 2005;49(4):275-80.
- [Background] Singh K, Gurha P. Comparative evaluation of Ambu AuraGain with ProSeal laryngeal mask airway in patients undergoing laparoscopic cholecystectomy. Indian J Anaesth. 2017 Jun;61(6):469-474. doi: 10.4103/ija.IJA_163_17. PMID 28655951
- [Background] Seet E, Rajeev S, Firoz T, Yousaf F, Wong J, Wong DT, Chung F. Safety and efficacy of laryngeal mask airway Supreme versus laryngeal mask airway ProSeal: a randomized controlled trial. Eur J Anaesthesiol. 2010 Jul;27(7):602-7. doi: 10.1097/eja.0b013e32833679e3. PMID 20540172
- [Background] 13. Soliman HF. Insertion characteristics of three supraglottic airway devices: A randomized comparative trial. Ain-Shams J Anaesthesiol. 2016;9(2):212-8.
- [Background] 14.Abdel-Halim TM, El Enin MA, Elgoushi MM, Afifi MG, Atwa HS. Comparative study between Air-Q and Intubating Laryngeal Mask Airway when used as conduit for fiber-optic. Egyptian J Anaesth. 2014;30(2):107-13.
- [Background] Brimacombe J, Keller C. The ProSeal laryngeal mask airway. Anesthesiol Clin North Am. 2002 Dec;20(4):871-91. doi: 10.1016/s0889-8537(02)00044-5. PMID 12512267
- [Background] Brimacombe J, Keller C, Boehler M, Puhringer F. Positive pressure ventilation with the ProSeal versus classic laryngeal mask airway: a randomized, crossover study of healthy female patients. Anesth Analg. 2001 Nov;93(5):1351-3, table of contents. doi: 10.1097/00000539-200111000-00064. PMID 11682428
- [Result] Galgon RE, Schroeder KM, Han S, Andrei A, Joffe AM. The air-Q((R)) intubating laryngeal airway vs the LMA-ProSeal(TM) : a prospective, randomised trial of airway seal pressure. Anaesthesia. 2011 Dec;66(12):1093-100. doi: 10.1111/j.1365-2044.2011.06863.x. Epub 2011 Aug 22. PMID 21880031
- [Result] Jagannathan N, Hajduk J, Sohn L, Huang A, Sawardekar A, Gebhardt ER, Johnson K, De Oliveira GS. A randomised comparison of the Ambu(R) AuraGain and the LMA(R) supreme in infants and children. Anaesthesia. 2016 Feb;71(2):205-12. doi: 10.1111/anae.13330. Epub 2015 Dec 9. PMID 26648173
- [Result] 4. Youssef MM, Lofty M, Hammad Y, Elmenshawy E. Comparative study between LMA-Proseal™ and Air-Q® Blocker for ventilation in adult eye trauma patients. Egyptian J Anaesth. 2014;30(3):227-33.
- [Result] 5. Sethi S, Maitra S, Saini V, Samara T. Comparison of Ambu® AuraGain™ laryngeal mask and air-Q™ intubating laryngeal airway for blind tracheal intubation in adults: a randomized controlled trial. Egyptian J Anaesthes. 2017;33(2):137-40.
- [Result] Joshi R, Rudingwa P, Kundra P, Panneerselvam S, Mishra SK. Comparision of Ambu AuraGain and LMA(R) ProSeal in children under controlled ventilation. Indian J Anaesth. 2018 Jun;62(6):455-460. doi: 10.4103/ija.IJA_86_18. PMID 29962528
- [Result] Brimacombe J, Keller C, Fullekrug B, Agro F, Rosenblatt W, Dierdorf SF, Garcia de Lucas E, Capdevilla X, Brimacombe N. A multicenter study comparing the ProSeal and Classic laryngeal mask airway in anesthetized, nonparalyzed patients. Anesthesiology. 2002 Feb;96(2):289-95. doi: 10.1097/00000542-200202000-00011. PMID 11818758
- [Result] Parikh DA, Jain RA, Lele SS, Tendolkar BA. A cohort evaluation of clinical use and performance characteristics of Ambu(R) AuraGain: A prospective observational study. Indian J Anaesth. 2017 Aug;61(8):636-642. doi: 10.4103/ija.IJA_285_17. PMID 28890558
- [Result] Wong DT, Ooi A, Singh KP, Dallaire A, Meliana V, Lau J, Chung F, Singh M, Wong J. Comparison of oropharyngeal leak pressure between the Ambu(R) AuraGain and the LMA(R) Supreme supraglottic airways: a randomized-controlled trial. Can J Anaesth. 2018 Jul;65(7):797-805. doi: 10.1007/s12630-018-1120-4. Epub 2018 Mar 26. PMID 29582360
- [Result] 11. Bhandari G, Mitra S, Shahi KS, Chand G, Tyagi A. A comparative study evaluating I-gel and Air-Q LMA for ventilation in anaesthetised and paralysed patients. Ann Int Med Dent Res. 2015;32:25-8.
- [Result] Lopez AM, Agusti M, Gambus P, Pons M, Anglada T, Valero R. A randomized comparison of the Ambu AuraGain versus the LMA supreme in patients undergoing gynaecologic laparoscopic surgery. J Clin Monit Comput. 2017 Dec;31(6):1255-1262. doi: 10.1007/s10877-016-9963-0. Epub 2016 Nov 26. PMID 27889843
- [Result] Darlong V, Biyani G, Pandey R, Baidya DK, Punj Ca. Comparison of performance and efficacy of air-Q intubating laryngeal airway and flexible laryngeal mask airway in anesthetized and paralyzed infants and children. Paediatr Anaesth. 2014 Oct;24(10):1066-71. doi: 10.1111/pan.12462. PMID 24961960
- [Result] 19. Lopez AM, Sala-Blanch X, Valero R, Prats A. Cross-over assessment of the AmbuAuraGain, LMA Supreme New Cuff and Intersurgical I-Gel in fresh cadavers. Open J Anesthesiol. 2014;4(12):332-9.